CLINICAL TRIAL: NCT01897129
Title: Human Papillomavirus and Pregnancy
Acronym: HPVandPregn
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ulla Bonde van Zwol (Other)
Collaborators: MCM Vaccines B.V. (Industry); Region of Southern Denmark (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Ulla Bonde van Zwol, MD, ph.d.-student, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: HPV AND PREGNANCY
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: HPV-infection in Pregnant Women

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biospecimen will be kept in a biobank for a period of 10 years after the end of this project. The biospecimens will be blood samples, cells collected from the ectocervix, vaginal microbioma, placental biopsies from prenatal diagnostics or miscarriages.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Early pregnancy: Women in early pregnancy at around the time of the nuchal translucency scan. The prevalence of HPV will be determined
- Chorionic villous sampling: Women undergoing chorionic villous sampling for the purpose of prenatal diagnostics.
- Spontaneous abortion: Women with miscarriage at a gestational age up to 22 weeks
- Preterm birth: Women with spontaneous preterm birth/premature primary rupture of membranes at a gestational age week 22-32
- Vaginal delivery at term: Women with spontaneous vaginal delivery at term (week 37+0-)
- Elective ceaserean section at term: Women undergoing elective cesarean section at term (week 37+0-)

SUMMARY:
Purpose Our study involves two hypotheses. One is that genital infection with HPV is associated with increased risk of miscarriage and preterm birth. The second hypothesis is that human papillomavirus can ascend from the vagina to the uterus through the cervix and cross the placental barrier. We wish to verify these hypotheses in our studies.

This study will determine the prevalence of HPV in Danish pregnant women and examine HPV's role in the aetiology of spontaneous abortion and preterm birth.

DETAILED DESCRIPTION:
Background Studies have shown significantly higher prevalence of HPV in tissue from miscarriages (60%) than from induced abortions (20%). HPV-infection in the extravillous trophoblasts in the placenta has furthermore been shown to induce cell death and cause dysfunction of the placenta, which can lead to adverse outcome of the pregnancy, e.g. preterm birth and hereby related neonatal mortality and morbidity. Spontaneous abortion and preterm birth are adverse events of the pregnancy, with for the biggest part unknown aetilogy, an area worth trying to elucidate by means of research.

Method 6 groups of each 91 women will be included:

* A group of early pregnant women at the nuchal translucency scan around gestational week 12 and a similar group undergoing chorion villous sampling in relation to prenatal diagnostics of the fetus
* A group of women with spontaneous abortion before gestational week 22 and a group with preterm birth gestational week 22-32
* A group delivering spontaneously at term and a group undergoing elective cesarean at term

The women will be examined by cervical swab to analyze for and do a genotyping of HPV if present. A vaginal swab will be done for the purpose of vaginal microbiome examination later. Furthermore analysis for HPV in placental tissue from chorion villous sampling or evacuation of the uterus after miscarriage. Cervical swabs and placental tissue will be analyzed by means of PCR (polymerase chain reaction) for the 35 types of HPV most frequently found in the anogenital area. Blood samples will be collected from all the patients and analyzed for HPV-antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women gestational week 10-42

Exclusion Criteria:

* Vaccinated against cervical cancer

Ages: 15 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women in Funen, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 546 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Human Papillomavirus infection of the uterine cervix in early pregnancy | 1st of November 2015
  Description of the prevalence of HPV in Danish pregnant women.

SECONDARY OUTCOMES:
Presence of Human Papillomavirus in uteri in the second trimester of pregnancy | 1st of November 2015
  Can HPV be found in the placenta during early pregnancy if the woman has HPV-infection on the ectocervix
Human Papillomavirus infection in the cervix uteri in pregnant women at term | 1st of November 2015
  The prevalence of HPV in Danish pregnant women at term

OTHER OUTCOMES:
HPV infection and preterm birth | 1st of November 2015
  Does HPV-infection in the cervix uteri increase the risk of preterm birth?
HPV infection and miscarriage | 1st of November 2015
  Does HPV infection increase the risk of miscarriage?

CONTACTS AND LOCATIONS:
Overall Officials: Jan S Joergensen, Doctor, Study Chair — Supervisor
Locations (1):
- Department of Gynecology and Obstetrics, Odense, Funen, Denmark